CLINICAL TRIAL: NCT03980106
Title: Comparing the Reciprocal Inhibition Method and Post-isometric Inhibition Method of Muscle Energy Technique on the Spinal Reflex Excitability in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of North Georgia (Other)
Responsible Party: Principal Investigator, Mohammad(Reza) Nourbakhsh, Professor of Physical Therapy, University of North Georgia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB 2019-026
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Relaxation; Joint; Limitation, Mobility; Relaxation; Lumbosacral
Keywords: Spinal Reflex Excitability; Muscle Relaxation; H reflex
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental RI-PI (Experimental): They receive the Reciprocal Inhibition (RI) technique in the first stage and then the Post-isometric Inhibition (PI) technique in the second stage.
  Interventions: Other: Reciprocal Inhibition Muscle Energy Technique; Other: Post-Isometric Inhibition Muscle Energy Technique
- Experimental PI-RI (Experimental): They receive the Post-isometric Inhibition (PI) technique in the first stage and then the Reciprocal Inhibition (RI) technique in the second stage.
  Interventions: Other: Reciprocal Inhibition Muscle Energy Technique; Other: Post-Isometric Inhibition Muscle Energy Technique

INTERVENTIONS:
Other: Reciprocal Inhibition Muscle Energy Technique — In this technique, the subject will be asked to contract antagonist muscles against a moderate resistant force provided by the therapist to inhibit the contraction of the agonist muscle.
Other: Post-Isometric Inhibition Muscle Energy Technique — In this technique, the subject will be asked to contract agonist muscles against a moderate resistant force provided by the therapist to inhibit the contraction of the agonist muscle.

SUMMARY:
This a cross-over study to compare the effect of two different muscle energy techniques (MET) including post-isometric inhibition and reciprocal inhibition on the spinal reflex excitability. The study contains two experimental groups, while one group will receive post-isometric inhibition MET in the first stage and reciprocal inhibition MET in the second stage, the other group will receive reciprocal inhibition MET in the first stage and post-isometric inhibition MET in the second stage.

DETAILED DESCRIPTION:
Reciprocal inhibition MET works based on the two mechanisms a) voluntary activation of agonist muscle that is simultaneously accompanied by the inhibition of the antagonist muscles or b) the activation of muscle spindle which causes a reflexive contraction in the agonist muscle (known as the stretch reflex) and relaxation of the antagonist muscles. By using this method, the activation of agonist muscles may inhibit or deactivate the antagonist muscles which may permit the therapist to introduce further ROM to the affected joint.

The other method of MET is post-isometric relaxation which works based on the two mechanisms including; 1) activation of Golgi Tendon Organs (GTO) that located between the muscle belly and its tendon and 2) presetting muscle spindles by muscle contraction witch project information to the spinal cord via afferent type II fibers and through a complex central control systems, the spindle is preset to adjust the tone of the muscle. It seems that moderate isometric contraction of muscle may preset the muscle spindle and cause a post-isometric relaxation within the agonist muscles which now can be stretched further, and this may permit the therapist to introduce further ROM to the affected joint and help to improve joint mobilization.

ELIGIBILITY:
Inclusion Criteria:

* without current low back pain

Exclusion Criteria:

* Suffering from pain in the cervical, thoracic and lumbar spine,
* Presenting signs of radiculopathy or peripheral neuropathy such as specific patterns of numbness and muscle weakness,
* Any history or signs of joint instability, healing fractures, malignancy, open wounds, sutures, severe rheumatoid arthritis.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-06 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in H Reflex Amplitude | First measurement (Base-line), second measurement after 30 minutes (Pre-test), third measurement after 20 minutes (first post-test), forth measurement after 20 minutes (second post-test)
  H reflex or Hoffman's reflex is a refectory reaction of muscles after electrical stimulation of sensory fibers (Ia afferent from muscle spindles) in their innervated nerves (here is Tibial N),
Change in M wave Amplitude | First measurement (Base-line), second measurement after 30 minutes (Pre-test), third measurement after 20 minutes (first post-test), forth measurement after 20 minutes (second post-test)
  M- wave is a compound muscle action potential, which is produce by the electrical stimulation of motor nerve fibers (here is Tibial N)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Nourbakhsh, Principal Investigator — Professor of Physical Therapy
Locations (1):
- University of North Georgia, Dahlonega, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
No Plan to share individual participant data to other researchers.